CLINICAL TRIAL: NCT03162393
Title: The Optimal Surgical Strategy for the Treatment of Total Brachial Plexus Avulsion Injury Patients
Brief Title: The Surgical Treatment of Total Brachial Plexus Avulsion Injury-A Retrospective Study of 73 Patients
Status: Completed | Type: Observational
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Kaiming Gao, Doctor, Huashan Hospital
Other Study IDs: NSFC-H0605/81501871
Record Dates: First submitted 2017-05-19; First posted 2017-05-22 (Actual); Last update posted 2017-05-22 (Actual); Status verified 2017-05

CONDITIONS: Brachial Plexus Injury
Keywords: brachial plexus; avulsion injury
MeSH Terms: conditions — Fractures, Avulsion | interventions — Nerve Transfer

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- group 1: phrenic nerve transfer to musculocutaneous nerve; spinal accessory transfer to suprascapular nerve; intercostal nerve transfer to triceps branch, radial nerve and axillary nerve; contralateral C7 nerve transfer to median nerve
  Interventions: Procedure: nerve transfer
- group 2: phrenic nerve transfer to musculocutaneous nerve; spinal accessory transfer to suprascapular nerve; intercostal nerve transfer to triceps branch and radial nerve; contralateral C7 nerve transfer to median nerve
  Interventions: Procedure: nerve transfer
- group 3: spinal accessory transfer to suprascapular nerve; intercostal nerve transfer to triceps branch, radial nerve and axillary nerve; contralateral C7 nerve transfer to median nerve and musculocutaneous nerve
  Interventions: Procedure: nerve transfer
- group 4: spinal accessory transfer to suprascapular nerve; intercostal nerve transfer to triceps branch and radial nerve; contralateral C7 nerve transfer to median nerve and musculocutaneous nerve
  Interventions: Procedure: nerve transfer
- group 5: spinal accessory transfer to suprascapular nerve; intercostal nerve transfer to musculocutaneous nerve, radial nerve and axillary nerve; contralateral C7 nerve transfer to median nerve and triceps branch
  Interventions: Procedure: nerve transfer
- group 6: spinal accessory transfer to suprascapular nerve; intercostal nerve transfer to musculocutaneous nerve and radial nerve; contralateral C7 nerve transfer to median nerve and triceps branch
  Interventions: Procedure: nerve transfer

INTERVENTIONS:
Procedure: nerve transfer

SUMMARY:
Brachial plexus avulsion injury (BPAI) caused by traction injury, especially total root avulsion, represents a severe handicap for the patient. Despite recent progress in diagnosis and microsurgical repair, the prognosis in such cases remains unfavorable. We need to find an relatively optimal surgical treatment.

DETAILED DESCRIPTION:
Brachial plexus avulsion injury (BPAI) caused by traction injury, especially total root avulsion, represents a severe handicap for the patient. Despite recent progress in diagnosis and microsurgical repair, the prognosis in such cases remains unfavorable. Nerve transfer is the most successful method for repairing cases of brachial plexus root avulsion. Phrenic nerve transfer, accessory nerve transfer, intercostal nerve transfer and contralateral C7 transfer are all well-established technique in the treatment of certain severe brachial plexus lesions in adults. As reported in previous articles, shoulder function, elbow flexion, elbow extension, and wrist and finger function have been restored successfully by spinal accessory, phrenic, intercostal, and contralateral C7 nerve transfers . However, the results of just one function reconstruction were evaluated in those articles. Few studies were found that focused on the whole function reconstructions of the affected limb. In different medical organizations even in our department, many different surgical strategies were used in treating total BPAI patients and the results differed significantly. Here, we investigated the results of different commonly used nerve transfer in order to determine a relatively optimal surgical strategy for treatment of total BPAI patients.

ELIGIBILITY:
Inclusion Criteria:

* global root avulsion brachial plexus injury, a minimum postoperative interval of 3 years, all operations performed by the same medical team, nerve transfer was the only reconstruction method.

Exclusion Criteria:

* diabetes, Volkmann contracture, fracture on the affected limb, rib fracture, brain trauma.

Ages: 12 Years to 60 Years | Sex: All
Age Groups: Child, Adult
Study Population: Between 1999 and 2006, a total of approximately 200 patients with posttraumatic total BPAI underwent surgical exploration and reconstruction of the brachial plexus and 109 agreed to participate in our study. Seventy-three patients were enrolled and 36 were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
physical examination | at least 3 years post-operative
  the motor and sensory function recovery of the recipient nerves